CLINICAL TRIAL: NCT03005340
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Pharmacokinetic Characteristics After Coadministration of C1-R215 and C2-R215 Compared to the Administration of C1-R215 and C2-R215 Independently in Healthy Male Volunteers
Brief Title: A Phase 1 Drug Drug Interaction Clinical Trial of C1-R215 and C2-R215 in Healthy Male Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Alvogen Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AK-CTR215-I-01
Record Dates: First submitted 2016-12-23; First posted 2016-12-29 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Healthy
MeSH Terms: interventions — bazedoxifene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group A (Active Comparator): Period 1: Bazedoxifene 20 mg Period 2: Cholecalciferol granule 10 mg Period 3: Bazedoxifene 20 mg+Cholecalciferol granule 10 mg
  Interventions: Drug: Treatment B; Drug: Treatment C; Drug: Treatment BC
- Group B (Active Comparator): Period 1: Bazedoxifene 20 mg Period 2: Bazedoxifene 20 mg+Cholecalciferol granule 10 mg Period 3: Cholecalciferol granule 10 mg
  Interventions: Drug: Treatment B; Drug: Treatment C; Drug: Treatment BC
- Group C (Active Comparator): Period 1: Cholecalciferol granule 10 mg Period 2: Bazedoxifene 20 mg Period 3: Bazedoxifene 20 mg+Cholecalciferol granule 10 mg
  Interventions: Drug: Treatment B; Drug: Treatment C; Drug: Treatment BC
- Group D (Active Comparator): Period 1: Cholecalciferol granule 10 mg Period 2: Bazedoxifene 20 mg+Cholecalciferol granule 10 mg Period 3: Bazedoxifene 20 mg
  Interventions: Drug: Treatment B; Drug: Treatment C; Drug: Treatment BC
- Group E (Active Comparator): Period 1: Bazedoxifene 20 mg+Cholecalciferol granule 10 mg Period 2: Cholecalciferol granule 10 mg Period 3: Bazedoxifene 20 mg
  Interventions: Drug: Treatment B; Drug: Treatment C; Drug: Treatment BC
- Group F (Active Comparator): Period 1: Bazedoxifene 20 mg+Cholecalciferol granule 10 mg Period 2: Bazedoxifene 20 mg Period 3: Cholecalciferol granule 10 mg
  Interventions: Drug: Treatment B; Drug: Treatment C; Drug: Treatment BC

INTERVENTIONS:
Drug: Treatment B — Bazedoxifene 20 mg
  Other Names: Bazedoxifene 20 mg
Drug: Treatment C — Cholecalciferol granule 10 mg
  Other Names: Cholecalciferol granule 10 mg
Drug: Treatment BC — Bazedoxifene 20 mg, Cholecalciferol granule 10 mg
  Other Names: Bazedoxifene 20 mg, Cholecalciferol granule 10 mg

SUMMARY:
Randomized, open-label, single-dose, three-treatment, six-sequence, three-way crossover study to evaluate the safety and pharmacokinetic characteristics after coadministration of C1-R215 and C2-R215 compared to the administration of C1-R215 and C2-R215 independently in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male between 19 and 45
* BW is above 50kg and BMI is between 18.5 and 30.0
* Subject who agreed and signed on informed consent form prior to the study participation

Exclusion Criteria:

* Presence or history of clinically significant disease
* Treatment history of any drug which might affect IP within 10days
* History of other study drugs within 12weeks

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-12; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve(AUCt) of Bazedoxifene | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120h
Area under the plasma concentration versus time curve(AUCt) of Cholecalciferol | -24, -12, -6, 0, 2, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 60, 72, 96h
Peak plasma concentration(Cmax) of Bazedoxifene | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120h
Peak plasma concentration(Cmax) of Cholecalciferol | -24, -12, -6, 0, 2, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 60, 72, 96h

CONTACTS AND LOCATIONS:
Overall Officials: Park, Principal Investigator — Dong-A University Hospital

IPD SHARING:
Plan to Share IPD: No